CLINICAL TRIAL: NCT00824187
Title: A Multicenter, Double-blind, Randomized, Placebo Controlled Study of the Monophasic Oral Contraceptive YAZ (20 µg Ethinylestradiol, 3 mg Drospirenone) in the Treatment of Chinese Patients With Premenstrual Dysphoric Disorder (PMDD)
Brief Title: YAZ Premenstrual Dysphoric Disorder (PMDD) in China
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Bayer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 91771; 311962 (Other: Company Internal)
Record Dates: First submitted 2009-01-15; First posted 2009-01-16 (Estimated); Last update posted 2014-04-02 (Estimated); Status verified 2014-04

CONDITIONS: Premenstrual Dysphoric Disorder ( PMDD)
Keywords: Premenstrual Dysphoric Disorder ( PMDD); Oral contraceptive
MeSH Terms: conditions — Premenstrual Dysphoric Disorder

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Arm 1 (Experimental)
  Interventions: Drug: EE20/DRSP(YAZ, BAY86-5300)
- Arm 2 (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: EE20/DRSP(YAZ, BAY86-5300) — 20 μg ethinylestradiol, 3mg drospirenone, tablet, orally, opd
  Arms: Arm 1
Drug: Placebo — Inert tablet
  Arms: Arm 2

SUMMARY:
The purpose of this study is to evaluate the efficacy and safety of YAZ compared to placebo in the treatment of symptoms related to Premenstrual Dysphoric Disorder (PMDD).

ELIGIBILITY:
Inclusion Criteria:

* Chinese women of reproductive age 18-45 years (inclusive) with a diagnosis of Premenstrual Dysphoric Disorder (PMDD)

Exclusion Criteria:

* Any formal psychotherapeutic counselling within 1 month before the screening visit (Visit 1) or used medication for Premenstrual Syndrome (PMS) or Premenstrual Dysphoric Disorder (PMDD) including, but not limited to hormones, bromocriptine, GnRH agonists, vitamin B6 (>100 mg), calcium supplements (> 1500 mg/day), anxiolytics and antidepressants during the 3 month period prior to Visit 1
* Use of sleeping medication (including melatonin) for more than 3 days per month.
* Pregnancy or less than 3 menstrual cycles since delivery, abortion or lactation before start of treatment
* Obesity (body mass index or BMI > 30 kg/m2)
* Hypersensitivity to any ingredient of the study drug

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 187 (Actual)
Dates: Start 2009-01; Primary Completion 2011-01 (Actual); Study Completion 2011-01 (Actual)

PRIMARY OUTCOMES:
The difference in DRSP scale scores for the first 21 items, comparing average scores from the last 5 days before menses of the 3rd cycle in the treatment phase to average scores from the last 5 days before menses of the 2 run in cycles | 3 cycles (1 cycle= 28 days)

SECONDARY OUTCOMES:
The difference in DRSP scale scores for the 3 functional impairment items, comparing the average over the last 5 days of daily scores from the 3rd cycle in the treatment phase to the average of daily scores from the 2 run in cycles | 3 cycles
Descriptive statistics for total DRSP scale scores (sum of the first 21 items) of the last 5 days for each of the 2 run in cycles, each of the 3 cycles in the treatment phase, and the average of the 3 cycles in the treatment phase | 3 cylces
Descriptive statistics for change in total DRSP scale scores (sum of the first 21 items) of the last 5 days from baseline to each cycle in the treatment phase and to the average of the 3 cycles in the treatment phase | 3 cycles
Assessment of CGI scores | 3 cycles
Adverse events | Whole study period
Laboratory tests | Whole study period

CONTACTS AND LOCATIONS:
Overall Officials: Bayer Study Director, Study Director — Bayer
Locations (12):
- China (12):
  - Guangzhou, Guangdong
  - Wuhan, Hubei
  - Changsha, Hunan
  - Nanjing, Jiangsu
  - Dalian, Liaoning
  - Jinan, Shandong
  - Xi’an, Shanxi
  - Chengdu, Sichuan
  - Kunming, Yunnan
  - Hangzhou, Zhejiang
  - Beijing
  - Tianjin